CLINICAL TRIAL: NCT04721327
Title: Remote Care: The Future of Cochlear Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Principal Investigator, Meredith Holcomb, Associate Professor, Director of Cochlear Implants, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20201410
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cochlear Implants
Keywords: telemedicine; service delivery model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Arm (Experimental): Patient ages 1-17 years who are current cochlear implant (CI) users will receive CI programming in person for the first visit and remotely for the second visit.
  Interventions: Other: remote CI programming
- Adult Arm (Experimental): Patient ages 18-90 years who are current cochlear implant (CI) users will receive CI programming in person for the first visit and remotely for the second visit.
  Interventions: Other: remote CI programming

INTERVENTIONS:
Other: remote CI programming — provision of CI programming provided remotely via Zoom in a 2 hour session

SUMMARY:
The purpose of this study is to see if remote programming visits for cochlear implants are possible.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Arm

1. English speaking patients (Parents can speak English and/or Spanish)
2. ages 1-17 years
3. current CI users with a Cochlear Americas device
4. minimum of 6-months of CI experience
5. maximum of 4 years of CI experience

Adult Arm

1. Postlingual patients
2. English speaking patients

2. ages 18-90 years 3. current CI users with a Cochlear Americas device 4. minimum of 3-months of CI experience 5. maximum of 18-months of CI experience

Exclusion Criteria:

1. Patients with physical neuropathy, abnormal anatomy (e.g., cochlear malformations), severe cognitive deficits, and/or severe mental health difficulties
2. Patients who do not speak English
3. Patients who do not have access to the internet
4. Patients who do not live in Florida
5. Patients who have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
electrode impedances | up to 8 months
  measured via CI programming software (kOhm)
electrically evoked compound potential values (neural response telemetry) | up to 8 months
  measured via CI programming software (mV)
datalogging | up to 8 months
  measured via CI programming software (hours per week)
stimulation levels | up to 8 months
  threshold and upper stimulation levels measured via CI programming software (clinical unit)
auditory skills as measured by the LittleEars Questionnaire | up to 8 months
  The LittleEars auditory questionnaire (LEAQ) uses parent responses to assess auditory behavior in children up to 24 months of age. The questionnaire is scored from 0 to 35 with 0 indicating poorer performance and 35 indicating better performance.
auditory skills as measured by the Auditory Skills Checklist (ASC) | up to 8 months
  ASC has a Total Score ranges from zero to 70, with higher scores indicating development of increasingly complex listening skills
hearing disability as measured by the Speech, Spatial and Qualities Hearing Scale (SSQ) | up to 8 months
  The SSQ is a a 49 item self-report test of hearing disability across three main sections and 10 pragmatic subscales. The total score ranges from zero to ten, with a lower score indicating a higher degree of hearing disability

SECONDARY OUTCOMES:
Behavior Assessment System for Children, 3rd Edition (BASC-3) | up to 8 months
  BASC-3 is scored 0-120 as a T score. Any scores between 60-70 is considered at risk / requires monitoring and scores greater than 70 are considered clinically significant / an area that likely requires therapeutic intervention.
Patient Health Questionnaire (PHQ-8) | up to 8 months
  PHQ-8 has 8 items rated on a scale from "not at all" (0) to "nearly every day" (3), with higher scores indicating greater frequency of depressive symptoms. The sum of the items indicates the overall level of depressive symptoms indicating mild (5-9), moderate (10-14), moderately severe (15-19), and severe depressive symptoms (20- 24).
Generalized Anxiety Disorder-7 (GAD-7) | up to 8 months
  GAD-7 is a 7-item self-report questionnaire of anxiety symptomatology in the past 14 days. Respondents rate the frequency of each item during the past two weeks on a 0-3-point scale ranging from not at all (0) to nearly every day (3). The sum of the items indicates the overall level of anxiety symptoms indicating mild (0-4), moderate (5-9), moderately severe (10-14), and severe (15- 21).
Quality of Life- CI (QoL-CI) | up to 8 months
  QoL-CI is scored 0-100 with higher scores indicating better quality of life.
Cochlear Implant Quality of Life-35 Profile (CIQOL-35 Profile) | up to 8 months
  CIQOL-35 Profile is a 35 item questionnaire with a total score ranging from 0-100% with a higher score indicating a higher level of functional ability with a cochlear implant
Parenting Stress Index/Short Form (PSI) | up to 8 months
  Parenting Stress Index/Short Form (PSI) contains 36 items rated on a 6-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree) and a total score. Higher scores indicate increased parenting stress.
Parenting Stress-CI | up to 8 months
  Parenting Stress-CI is completed by the parent and scored from "not at all stressful" (0) to "very stressful" (3) with higher scores indicating greater degrees of parenting stress. For parents of children 0-5 years, there are 15 items. For parents of children 6-12 years there are 8 items.
Scale of Parental Involvement and Self-Efficacy-Revised (SPISE-R) | up to 8 months
  The SPISE-R is comprised of 46 questions that uses a 7-point Likert scale to query parents' beliefs, knowledge, confidence, and actions relevant to supporting their child's auditory access and spoken language development. The total average score will range from 1 to 7 with 7 indicating the highest score / highest level of parental involvement and self efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Holcomb, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No